CLINICAL TRIAL: NCT02704234
Title: Acupuncture for Vulvodynia: A Double-blinded Feasibility Pre-pilot Study
Brief Title: Acupuncture for Vulvodynia: A Pre-pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Judith Schlaeger, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015-0692
Record Dates: First submitted 2015-11-30; First posted 2016-03-09 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Vulvodynia; Vulvar Vestibulitis; Dyspareunia; Pain
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis; Dyspareunia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Acupuncture (Experimental): Active Acupuncture 2 times per week for 5 weeks
  Interventions: Other: Active Acupuncture
- Placebo (Placebo Comparator): Placebo Acupuncture 2 times per week for 5 weeks
  Interventions: Other: Placebo Acupuncture

INTERVENTIONS:
Other: Active Acupuncture — Active Acupuncture two times per week for 5 weeks
  Other Names: Penetrating Acupuncture Needle
  Arms: Active Acupuncture
Other: Placebo Acupuncture — Placebo Acupuncture two times per week for 5 weeks
  Arms: Placebo

SUMMARY:
Vulvodynia is a women's pain condition. Women have pain in their vulva, the area in their genitals between the vagina and labia (lips of the vagina). They also have pain when they have sexual intercourse or insert anything in the vagina. Sometimes they have so much pain, that they cannot have sex.

This research is being done for two reasons. The first reason is to test a set of special needles called double-blinded acupuncture needles to give acupuncture treatments (one is a real needle and the other is a fake needle). The second reason is to develop a protocol (checklist) that will be used in this and future studies, and to identify and resolve any procedural problems. The protocol will be first tested by the principal investigator who is also an acupuncturist. The investigator will perform acupuncture using the protocol, if necessary change the protocol, and then teach a second acupuncturist using the modified protocol how to use the double-blinded acupuncture needles.

The real needle called the penetrating needle penetrates the skin. The fake needle called the non-penetrating placebo touch needle does not penetrate the skin but it touches the skin so it feels like a needle is being inserted. It has a blunt tip.

Participants can't see which needle they are getting acupuncture with because the needles are housed in a double-blinded needle device which has two tubes (an inner and an outer) that neither the acupuncturists nor the participants can see through.

If a fake acupuncture needle can be used in acupuncture research like a sugar pill is used for drug studies to see how well the real medicine works, the investigators can see how effective acupuncture is. The investigators will be testing these needles to treat participants with vulvodynia.

ELIGIBILITY:
Inclusion Criteria:

* women previously diagnosed with generalized vulvodynia
* women previously diagnosed with localized vestibulodynia,

Exclusion Criteria:

* pregnancy
* menopause
* interstitial cystitis
* irritable bowel syndrome
* untreated vaginitis
* cervicitis
* pelvic inflammatory disease
* any other pelvic pathology causing pain
* concomitant physical therapy
* concomitant biofeedback
* concomitant massage
* additional acupuncture

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Change in Vulvar Pain Scale | baseline and twice weekly for 5 weeks
  PainReportIt, the computerized McGill Pain Questionnaire
Change in Dyspareunia Questionnaire | baseline and once per week for 5 weeks
  Female Sexual Function Index

SECONDARY OUTCOMES:
Vulvar Function Status Questionnaire | at baseline and 5 weeks
  Assesses vulvar function

OTHER OUTCOMES:
Sleep Quality Scale | at baseline and 5 weeks
  Pittsburgh Sleep Quality Index
The Protocol Acceptability Scale for Treating Vulvodynia with Acupuncture | 5 weeks
  Acceptability of the acupuncture protocol for the participant
Double-Blinded Needle Questionnaires for the Acupuncturist and for the Participant | 5 weeks
  Assesses the Ability of the Acupuncturist and Subject to Remain Blind

CONTACTS AND LOCATIONS:
Overall Officials: judith schlaeger, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- A Center for Oriental Medicine, Wilmette, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schlaeger JM, Takakura N, Yajima H, Takayama M, Steffen AD, Gabzdyl EM, Nisi RA, McGowan Gruber K, Bussell JM, Wilkie DJ. Double-blind acupuncture needles: a multi-needle, multi-session randomized feasibility study. Pilot Feasibility Stud. 2018 Apr 13;4:72. doi: 10.1186/s40814-018-0265-9. eCollection 2018. PMID 29686883